CLINICAL TRIAL: NCT03307161
Title: Osteopathic Manual Treatment of Postural Abnormality, Pain, and Autonomic Control of Cardiac Function in People With Parkinson's Disease and Truncal Dystonia
Brief Title: Osteopathic Manual Treatment Parkinson's Disease and Truncal Dystonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1130
Record Dates: First submitted 2017-10-06; First posted 2017-10-11 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease; Dystonia; Autonomic Dysreflexia
Keywords: manual therapy; heart rate
MeSH Terms: conditions — Parkinson Disease; Dystonia; Autonomic Dysreflexia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Parkinsons fwd posture manual treatment (Active Comparator): Subject will receive the intervention, osteopathic manual treatment protocol.
  Interventions: Other: osteopathic manual therapy
- Parkinsons forward posture (No Intervention): Subjects will receive counseling.
- Parkinsons without forward posture (No Intervention): Subjects will receive counseling.

INTERVENTIONS:
Other: osteopathic manual therapy — Investigators board certified in osteopathic manual therapy will use their hands in a non-invasive manner to improve dystonia symptoms
  Arms: Parkinsons fwd posture manual treatment

SUMMARY:
This study will determine if posture and heart rate variability will significantly improve in Parkinsons disease with camptocormia after osteopathic manual treatments dystonia.

DETAILED DESCRIPTION:
This study will determine if posture and heart rate variability will significantly improve in Parkinsons disease with camptocormia after receiving 8-weekly sessions of the osteopathic manual treatments for truncal flexion dystonia as measured by the distance of the external acoustic meatus from a plumb-line to lateral malleolus, spinal X ray, and heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease; able to stand for three minutes or more

Exclusion Criteria:

* severe dementia, moderate or severe hallucinations and psychosis; unable to stand for three minutes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11; Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
change in posture | 8 weeks
  inches of forward head carriage
change in heart rate variability | 8 weeks
  heart rate changes

CONTACTS AND LOCATIONS:
Overall Officials: Jayme Mancini, PhD DO, Principal Investigator — NYIT col osteopathic medicine
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No